CLINICAL TRIAL: NCT05108415
Title: Blood Specimen Collection Study for NAFLD
Brief Title: Development and Validation of a Multi-target, Blood-based NAFLD Diagnosis Test
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: HBI Solutions Inc. (Industry)
Collaborators: mProbe Inc. (Industry)
Responsible Party: Principal Investigator, James Shilling, Principal Investigator, HBI Solutions Inc.
Other Study IDs: NAFLD_001
Record Dates: First submitted 2021-10-25; First posted 2021-11-05 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: NAFLD; NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort A: Blood specimen collection.
  Study samples must be collected prior to any treatment.
- Cohort B: Blood specimen collection.
  Samples must be collected prior to perform the ultrasonography.
- Cohort C: Blood specimen collection.
  Study samples must be collected prior to any treatment.

SUMMARY:
Multi-omics approach was used to identify patterns of serological biomarkers to diagnose NAFLD. The purpose of this study is to develop and validate a blood-based assay to diagnose NAFLD by collecting blood sample from healthy patients undergoing routine screening ultrasonography and from patients recently diagnosed with NAFLD.

DETAILED DESCRIPTION:
Accurate diagnosis of NAFLD combined with effective treatment improves survival and quality of life. Multi-omics approach was used to identify patterns of serological biomarkers to diagnose NAFLD. The purpose of this study is to develop and validate a blood-based assay for accurate diagnosis of NAFLD. The study will collect blood sample from healthy patients undergoing routine screening ultrasonography and from patients recently diagnosed with NAFLD. A blood-based test for NAFLD could offer an accurate, convenient, and patient-friendly screening option for current and future generations, and, in doing so, could save and improve lives by increasing adherence and accurate diagnosis.

Three types of patients in this study:

Cohort A:

People ages 20-85 who have been recently diagnosed with (or strong clinical suspicion for) NAFLD. Blood samples must be collected before any treatment has been initiated.

Cohort B:

People ages 20-85 undergoing routine screening ultrasonography for NAFLD as part of their regular medical check-ups. Blood samples must be collected before ultrasonography.

Cohort C:

People ages 20-85 who have been recently diagnosed with (or strong clinical suspicion for) NASH, an extremely advanced form of non-alcoholic fatty liver disease (NAFLD), is defined as hepatic steatosis with inflammation and hepatocyte injury. Blood samples must be collected before any treatment has been initiated.

ELIGIBILITY:
COHORT A

Inclusion Criteria:

* 20-85 years of age
* Recently completed ultrasonography examination.
* Recently diagnosed with (or strong clinical suspicion for) primary NAFLD.
* At least 7 days before but no more than 2 months after the most recent ultrasonography
* Able and willing to provide blood samples per protocol
* Able to comprehend and willing to sign and date the written informed consent document(s) and any applicable medical record release documents for the study

Exclusion Criteria:

* Alcohol abuse (weekly ethanol consumption: >140 g for men and >70 g for women) in the past year.
* Personal history of NAFLD (other than most recent diagnosis)
* Ultrasonography within the previous 9 years (other than most recent diagnosis)
* A history of fatty liver or other liver diseases such as autoimmune hepatitis and drug-induced liver disease.
* Have a medical condition which, in the opinion of the investigator, should preclude enrollment into the study.
* Have participated or be currently participating in a clinical research study in which an experimental medication has been administered during the 60 days up to and including the date of providing informed consent or may be administered through the time of the ultrasonography.
* If female, known to be pregnant.

COHORT B

Inclusion Criteria:

* 20-85 years of age
* Planning to undergo a screening ultrasonography within 2 months after providing signed informed consent
* Able and willing to provide blood samples per protocol
* Able to comprehend and willing to sign and date the written informed consent document(s) and any applicable medical record release documents for the study

Exclusion Criteria:

* Alcohol abuse (weekly ethanol consumption: >140 g for men and >70 g for women) in the past year.
* Personal history of NAFLD
* Ultrasonography within the previous 9 years
* A history of fatty liver or other liver diseases such as autoimmune hepatitis and drug-induced liver disease.
* Have a medical condition which, in the opinion of the investigator, should preclude enrollment into the study.
* Have participated or be currently participating in a clinical research study in which an experimental medication has been administered during the 60 days up to and including the date of providing informed consent or may be administered through the time of the ultrasonography.
* If female, known to be pregnant.

COHORT C

Inclusion Criteria:

* 20-85 years of age
* Recently completed ultrasonography examination.
* Recently diagnosed with (or strong clinical suspicion for) NASH, an extremely advanced form of non-alcoholic fatty liver disease (NAFLD), defined as hepatic steatosis with inflammation and hepatocyte injury..
* At least 7 days before but no more than 2 months after the most recent ultrasonography
* Able and willing to provide blood samples per protocol
* Able to comprehend and willing to sign and date the written informed consent document(s) and any applicable medical record release documents for the study

Exclusion Criteria:

* Alcohol abuse (weekly ethanol consumption: >140 g for men and >70 g for women) in the past year.
* Personal history of NAFLD or NASH (other than most recent diagnosis)
* Ultrasonography within the previous 9 years (other than most recent diagnosis)
* A history of fatty liver or other liver diseases such as autoimmune hepatitis and drug-induced liver disease.
* Have a medical condition which, in the opinion of the investigator, should preclude enrollment into the study.
* Have participated or be currently participating in a clinical research study in which an experimental medication has been administered during the 60 days up to and including the date of providing informed consent or may be administered through the time of the ultrasonography.
* If female, known to be pregnant.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Confirmative of Number of Participants with NAFLD Diagnosis | 2 months
  Confirmative of number of Participants with NAFLD diagnosis in patients undergoing routine screening ultrasonography, or post-ultrasonography.

IPD SHARING:
Plan to Share IPD: Undecided